CLINICAL TRIAL: NCT00056498
Title: Clozapine Treatment of Schizophrenic Patients
Brief Title: Risperidone Treatment in Schizophrenia Patients Who Are Currently Taking Clozapine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Robert Buchanan, Professor of Psychiatry, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01 MH045074 H-21270; R01MH045074 (NIH); DSIR 83-ATAP
Record Dates: First submitted 2003-03-14; First posted 2003-03-17 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Participants assigned to risperidone
  Interventions: Drug: Risperdal
- Placebo (Placebo Comparator): Participants assigned to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo capsule daily for 16 weeks
  Arms: Placebo
Drug: Risperdal — Risperdal 4 mg per day for 16 weeks
  Other Names: Risperidone
  Arms: Active

SUMMARY:
This study will determine whether adding the drug risperidone (Risperdal®) is more effective than placebo in treating schizophrenic patients who are taking the drug clozapine.

DETAILED DESCRIPTION:
Clozapine is the only antipsychotic drug that has been approved for treatment resistant patients with schizophrenia. However, up to 50% of patients treated with clozapine fail to respond and continue to exhibit clinically significant residual positive and negative symptoms and cognitive impairments. An emerging trend in treatment is the addition of a second antipsychotic drug. This study will determine if risperidone when given as adjunctive treatment is more effective than placebo in treating schizophrenic patients failing clozapine therapy.

Participants are randomly assigned to add either adjunctive risperidone or placebo to their current clozapine treatment in a single, daily dose for 16 weeks. Positive and negative symptoms, cognitive impairments, side effects of the treatment, anxiety, depression, hostility symptoms, and quality of life are assessed. Neurological tests, self administered questionnaires, and interviews are used to assess patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for schizophrenia or schizoaffective disorder
* Current clozapine treatment
* Moderate illness severity and inadequate positive symptom response to clozapine treatment
* 6 month period of clozapine treatment with documented clozapine blood level greater than or equal to 350 ng/ml or clozapine and norclozapine blood level greater than or equal to 450 ng/ml

Exclusion Criteria:

* Organic brain disorder
* Mental retardation
* Medical condition whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
* Pregnancy
* DSM-IV criteria for current alcohol or substance dependence within the last 6 months or DSM-IV criteria for alcohol or substance abuse within the last month
* Previously received adjunctive risperidone (at doses greater than or equal to 8 mg/day) with their clozapine treatment for greater than or equal to 6 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2001-12 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- [Derived] Weiner E, Conley RR, Ball MP, Feldman S, Gold JM, Kelly DL, Wonodi I, McMahon RP, Buchanan RW. Adjunctive risperidone for partially responsive people with schizophrenia treated with clozapine. Neuropsychopharmacology. 2010 Oct;35(11):2274-83. doi: 10.1038/npp.2010.101. Epub 2010 Jul 21. PMID 20664583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Though funding was in place beginning in 2001, recruitment took place from 2003 to 2008. Subjects were recruited from the Maryland Psychiatric Research Center Outpatient Reseach clinic, the Treatment Research Program, and community mental health centers.
Pre-assignment Details: 86 Participants signed informed consent. 15 were ineligible or excluded. 71 Participants entered the evaluation phase. Two were withdrawn prior to randomization. Four people withdrew after randomization but prior to starting study medications.
Groups:
- Risperidone: Participants assigned to risperidone
Period: Overall Study
Arm/Group | Risperidone | Placebo
Started | 30 | 35
Completed | 25 | 28
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone | Placebo | Total
Number analyzed (Participants) | 30 | 35 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (7.2) | 44.1 (9.3) | 46.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 19 | 25 | 44
Region of Enrollment [Number; unit: participants]
  United States | 30 | 35 | 65.0

OUTCOME MEASURES:

1. Primary Outcome: Positive Symptom Item Scores by Week and Treatment Group
Description: The Brief Psychiatric Rating Scale (BPRS) positive symptom items are: conceptual disorganization, hallucinatory behavior, unusual thought content, and suspiciousness. The total score is calculated by adding the scores for each item. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum score is 4 and the maximum score is 28. A higher score indicates a more severe positive symptom rating. A mixed model for unbalanced repeated measures analysis of covariance (ANCOVA), in which follow-up symptom score = baseline symptom score + treatment + week + treatment x week, and week is treated as a categorical, rather than a continuous measure. The treatment term estimates the average across weeks of the week-specific group differences, and is used as the main test for treatment effects on symptom change.
Time Frame: Baseline and every two weeks for 16 weeks.
Population: The intent to treat analysis included all participants who received at least one dose of study medication and completed the BPRS rating at the specified week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Placebo
Number analyzed (Participants) | 30 | 34
units on a scale
  Week 0 | 15.5 (3.8) | 15.5 (4.2)
  Week 2 | 14.6 (3.7) | 15.1 (4.0)
  Week 4: number analyzed (Participants) | 28 | 34
  Week 4 | 13.3 (4.0) | 14.4 (3.5)
  Week 6: number analyzed (Participants) | 28 | 33
  Week 6 | 13.9 (3.9) | 14.7 (3.8)
  Week 8: number analyzed (Participants) | 28 | 33
  Week 8 | 13.5 (4.2) | 14.9 (3.9)
  Week 10: number analyzed (Participants) | 26 | 31
  Week 10 | 13.9 (4.2) | 14.9 (4.2)
  Week 12: number analyzed (Participants) | 25 | 31
  Week 12 | 13.8 (3.7) | 15.3 (4.6)
  Week 14: number analyzed (Participants) | 24 | 28
  Week 14 | 13.4 (3.5) | 14.2 (3.8)
  Week 16: number analyzed (Participants) | 25 | 28
  Week 16 | 13.2 (3.5) | 14.1 (3.6)
  Change Score | -2.6 (3.1) | -1.5 (3.4)

2. Secondary Outcome: Neuropsychological Testing - Overall Composite Z-score
Description: The neuropsychological testing measured attention, executive function/problem solving, motor speed, processing speed/response generation, and verbal, visual, and working memory. The individual test raw scores were converted to z-scores and an overall composite z-score was computed from the average of the individual test z-scores. Z-scores range from -3 standard deviations up to +3 standard deviations. Higher scores indicate better test performance.
Time Frame: Baseline and Week 16
Population: Two participants completed 9 or fewer of the 13 individual tests in the neurocognitive battery, and were omitted from calculation of the overall composite score
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Risperidone | Placebo
Number analyzed (Participants) | 24 | 27
z-score
  Baseline | 0.02 (0.66) | -0.03 (0.46)
  Week 16 | 0.12 (0.66) | 0.07 (0.47)

3. Secondary Outcome: Negative Symptom Total Score by Week and Treatment Group
Description: The Scale for the Assessment of Negative Symptoms (SANS) total score, minus the global items, inappropriate affect, poverty of content of speech, and attention items, used to measure negative symptoms. SANS total score range = 0-85. Higher scores indicate more severe negative symptoms. A mixed model for unbalanced repeated measures analysis of covariance (ANCOVA), in which follow-up symptom score = baseline symptom score + treatment + week + treatment x week, and week is treated as a categorical, rather than a continuous measure. The treatment term estimates the average across weeks of the week-specific group differences, and is used as the main test for treatment effects on symptom change.
Time Frame: Baseline and every two weeks for 16 weeks.
Population: The intent to treat analysis included all participants who received at least one dose of study medication and completed the SANS rating at the specified treatment week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Placebo
Number analyzed (Participants) | 30 | 34
units on a scale
  Week 0 | 32.3 (11.6) | 33.0 (13.3)
  Week 2 | 30.8 (11.5) | 34.0 (12.1)
  Week 4: number analyzed (Participants) | 28 | 34
  Week 4 | 29.8 (11.6) | 32.9 (13.3)
  Week 6: number analyzed (Participants) | 28 | 33
  Week 6 | 31.2 (10.3) | 33.0 (12.7)
  Week 8: number analyzed (Participants) | 27 | 33
  Week 8 | 30.4 (11.3) | 34.0 (14.1)
  Week 10: number analyzed (Participants) | 25 | 31
  Week 10 | 30.6 (10.9) | 33.1 (13.3)
  Week 12: number analyzed (Participants) | 25 | 31
  Week 12 | 31.6 (10.7) | 32.4 (12.5)
  Week 14: number analyzed (Participants) | 24 | 28
  Week 14 | 31.7 (11.0) | 34.4 (14.1)
  Week 16: number analyzed (Participants) | 25 | 28
  Week 16 | 31.3 (11.9) | 34.4 (14.8)
  Change Score | -2.6 (5.6) | 1.1 (10.8)

ADVERSE EVENTS:
Arm/Group | Risperidone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/35
Other Adverse Events (participants affected / at risk) | 0/30 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=30) | Placebo (N=35)
increased auditory hallucinations (Psychiatric disorders) | 1 | 0 — Participant was hospitalized due to an increase in intensity of auditory hallucinations including commands to harm self and need for hospitalization. Considered to be moderate in severity, and remotely study drug and concomitant drug related.
gastrointestinal symptoms (Gastrointestinal disorders) | 0 | 1 — Subject c/o of diarrhea, nausea, and vomiting with a history of constipation and admitted to the hospital. Subject was treated for renal failure secondary to nausea and vomiting. Considered to be severe and possibly drug related.
Panic attack (Psychiatric disorders) | 0 | 1 — Subject reported to the ER c/o racing pulse and thoughts and experiencing a "panic attack". After overnight observation, patient reports symptoms subsided and all labwork was normal. Determined to be severe and remotely study drug related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No